CLINICAL TRIAL: NCT01787084
Title: Transcatheter Valve Therapy (TVT) Registry Assessment of Alternative Access Approaches for Transcatheter Aortic Valve Replacement (TAVR) in Inoperable Patients With Severe Aortic Stenosis
Brief Title: Alternative Access Approaches for Transcatheter Aortic Valve Replace (TAVR) in Inoperable Patients With Aortic Stenosis
Acronym: Inop AA
Status: Completed | Type: Observational
Sponsor: The Society of Thoracic Surgeons (Other)
Collaborators: American College of Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: TVTR-2012-02
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Severe Symptomatic Aortic Stenosis
Keywords: Aortic Stenosis; TAVR
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inoperable Patients Alternative Access: Non-femoral delivery (or alternative access) in patients iwht severe symptomatic native aortic valve stenosis who have been determined by a cardiac surgeon to be inoperable for open aortic valve replacement and in whom existing co-morbidities would not preclude the expected benefit from correction of the aortic stenosis
  Interventions: Device: Edwards SAPIEN Transcatheter Heart Valve

INTERVENTIONS:
Device: Edwards SAPIEN Transcatheter Heart Valve — Non-femoral transcatheter delivery of heart valve

SUMMARY:
Investigational study of Edwards Lifesciences, LLC's "Edwards SAPIEN Transcatheter Heart Valve" for non-femoral delivery, (or alternative access deliver) in patients with severe symptomatic native aortic valve stenosis who have been determined by a cardiac surgeon to be inoperable for open aortic valve replacement and in whom existing co-morbidities would not preclude the expected benefit from correction of the aortic stenosis. Will outcomes observed in a high-risk operable transapical native valve TAVR cohort receiving an Edwards SAPIEN device compare to inoperable patients undergoing alternative access TAVR with the Edwards SAPIEN device experience a reasonably similar incidence of 30 day adverse events?

DETAILED DESCRIPTION:
Transcatheter aortic valve replacement (TAVR) using the Edwards SAPIEN valve and Retroflex 3 delivery system provides both a mortality and quality of life benefit for inoperable patients. Only the transfemoral (TF) access has been approved in the US. A substantial number of patients cannot have a TF approach due to inadequate vessel size, vessel disease, or other anatomical considerations. The pivotal study did not include an assessment of safety and effectiveness of alternative access approaches in this inoperable patient group.

Early approaches to TAVR included a femoral transvenous approach with transseptal access to the left side for delivery of the valve. This approach avoided large bore arterial catheterization, but it had unacceptable rates of complications and lacked reproducibility. Alternative access approaches have been developed because of the risks associated with inserting large caliber catheters into small, diseased femoral arteries often associated with diffuse vasculopathy. To avoid the vascular complications from femoral access, other transcatheter approaches have been developed to include open surgical access to the left ventricular apex (TA), ascending aorta, (TAO), subclavian and axillary arteries (TS), and retroperitoneal access to the iliac artery (TI) as well as distal aorta. In addition to providing TAVR to patients who cannot have TF access, additional advantages include better catheter control and safer closure of the access site. Commonly cited disadvantages include the need for surgical expertise and additional equipment, along with the potential for longer recovery, more incisional pain, greater radiation exposure for operators, unsuitable delivery catheters for alternative access sites, and a host of unique alternative access site complications.

We propose to collectively analyze 30-day safety endpoints as a lumped data group for these alternative access approaches. These data are gathered from clinical practice in real-world settings and submitted to the TVT Registry. It is expected that centers will choose among the various choices for alternative access based the causative factors underlying the need for alternative access, as well as local skill sets and experience. For this lumped data group of alternative access approaches we will compare 30-day safety results to the TA outcomes reported from Cohort A of the PARTNERS 1 trial. We recognize that these TA patients were high risk operable patients rather than inoperable patients, but no other direct comparator group is available. We reason that the TA data from this published clinical trial are high quality, represent an alternative access approach rather than TF, and will provide a frequency of safety endpoints that have been found to be acceptable both clinically and from a regulatory perspective.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Primary indication is symptomatic primary severe aortic stenosis predicted to benefit from relief of valvular stenosis
* Aortic valve area less than 0.8 centimeters squared
* Mean aortic valve gradient greater than or equal to 40 mmHG
* Peak aortic jet velocity greater than or equal to 4.0 m per second
* Valve sheath access site is femoral, axillary, transapical, transaortic, subclavian or subaxillary
* Patient is judged by the local heart team to be inoperable for Aortic Valve Replacement due to severe chest wall deformities or radiation effects, severe peripheral or aortic vascular disease, or severe systemic disease prohibiting the safe conduct of Cardiopulmonary Bypass (CPB)

Exclusion Criteria:

* Aortic valve annulus size is less than 18 mm or greater than 25 mm
* Active infectious endocarditis
* Valve in prosthetic valve procedure
* Patients considered by the heart team to be unlikely to receive meaningful or durable clinical benefit from the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will include all TVT Registry data obtained for inoperable patients age 18 years or older who undergo TAVR for severe aortic stenosis using any non-femoral access approach with an Edwards SAPIEN device between the start date and December 31, 2018
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-04; Primary Completion 2025-03 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events | 30 day
  Increase in the 30-day risk of adverse events among patients receiving TAVR; Modified 30 day Valve Academic Research Consortium (VARC) Composite Early Safety Endpoint
Mortality | 1 year
  Proportion of patients who are alive with at least moderate functional improvement (defined as at least 10 point improvement in Kansas City Cardiomyopathy Questionnaire (KCCQ) from baseline) at 1 year after TAVR

SECONDARY OUTCOMES:
30-day endpoints for major morbidity | 30 day
  Endpoints include: mortality, stroke, stroke or transient ischemic attack (TIA), major vascular complications, valve-related dysfunction requiring re-intervention, incident renal replacement therapy, life-threatening bleeding, and high-degree aortic valve (AV) block requiring permanent pacemaker implantation

CONTACTS AND LOCATIONS:
Overall Officials: John D Carroll, MD, Principal Investigator — American College of Cardiology; Fred H Edwards, MD, Principal Investigator — Society of Thoracic Surgeons